CLINICAL TRIAL: NCT03847129
Title: Functional Measurements and Therapeutic Intervention for Hand Neuropathy in Diabetes Mellitus
Brief Title: Assessments and Interventions for Hand Neuropathy in DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: B-ER-103-328
Record Dates: First submitted 2019-02-12; First posted 2019-02-20 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Diabetes Mellitus; Neuropathy, Diabetic
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Neuropathies | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Biofeedback training group (Experimental): The participants in the biofeedback training group attend a 30 minute biofeedback protocol per session, two times a week for six to eight weeks that is also combined with the regular diabetic care treatment in the Occupational Therapy Room.
  Interventions: Other: Biofeedback training
- Home-based training group (Active Comparator): The participants in this group receive similar doses of home-based tendon gliding exercises and resistance training with an anti-stress ball for 30 minutes at a frequency of 2 times a week for 6 to 8 weeks, also combined with the regular diabetic care treatment.
  Interventions: Other: Home-based tendon gliding and resistance training
- Control group (No Intervention): The participants in the control group receive only diabetes disease prevention consultation once and outcome assessments twice.

INTERVENTIONS:
Other: Biofeedback training — Before the biofeedback training, the baseline pinch force detected from a pinch-holding-up activity is recorded to set the target level according to the baseline data. With the aim for improving the performance, a 94% peak force value detected at the baseline is set as the target threshold for the training. Each participant attends a 30-minute biofeedback protocol per session, two times a week for six to eight weeks. Once the pinch force value exceeds the target range, visual and auditory cues are provided to inform the subjects to modify the performance.
  Arms: Biofeedback training group
Other: Home-based tendon gliding and resistance training — The participants receive similar doses of home-based tendon gliding exercises and resistance training with an anti-stress ball for 30 minutes at a frequency of 2 times a week for 6 to 8 weeks, also combined with the regular diabetic care treatment. Six to eight telephone visits are carried out to remind the patients to comply with the exercise program during the training period.
  Arms: Home-based training group

SUMMARY:
This study is to investigate the effects of task-based biofeedback training compared with home-based programs on sensorimotor function and quality of life for diabetic patients with neuropathic hands. The investigators hypothesize that the task-based biofeedback training might have significant effectiveness for restoration of sensory function, precision pinch performance, hand dexterity and life quality for patients with diabetic neuropathy.

DETAILED DESCRIPTION:
Hand tendon gliding exercises allow both the flexor digitorum profundus and superficialis tendons of hands to achieve the greatest range of motion. Thus, in conjunction with resistive exercises for diabetic hands, such exercises are considered an appropriate home-based training method that has positive effects on various diabetic hand problems in terms of regaining smooth tendon excursion, preventing joint contracture, and reducing intrinsic muscle tightness. Different from the biomechanical approach to deal with hand problems, a biofeedback system can be used to provide real-time information on improper movements during task-based training intended to enhance either performance quality or accuracy. This study aims to analyze the difference in treatment effects between a computerized evaluation and a re-education biofeedback system that provides interactive sensorimotor information to shape the optimized coordinated pinch pattern of a hand and a home-based tendon gliding exercise program in conjunction with resistive exercise with weekly supervision on sensorimotor function and quality of life for diabetic patients. The investigators hypothesize the task-based biofeedback training using the biofeedback training system could have significant effectiveness for restoration of sensory function, precision pinch performance, hand dexterity and life quality for patients with diabetic neuropathy.

ELIGIBILITY:
Inclusion Criteria:(for training groups)

* with clinically-defined type II DM who were diagnosed based on the 1997 American Diabetes Association criteria
* impaired in terms of force modulation in precision pinch performance as detected using the PHUA test are referred from outpatients from the Department of Family Medicine in a medical center in southern Taiwan

Exclusion Criteria:(for training groups and healthy control group)

* diagnosed neuro-musculoskeletal disorders
* traumatic nerve injuries of the upper limbs
* trauma to the hand or congenital anomalies of the wrist and hand
* skin infections or disease of the hands
* cognitive deficits
* aged less than 20 years old

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-08-20 (Actual); Primary Completion 2016-06-02 (Actual); Study Completion 2016-06-02 (Actual)

PRIMARY OUTCOMES:
The pinch-holding-up activity (PHUA) test | Baseline
  For the PHUA test, the participants were asked to pinch and lift the pinch device, and the pinch force will be recorded during the task. The raw force value would be collected and transferred into specific parameters include: (1) FP_Peak: the maximum pinch force during the lifting phase in the PHUA test; (2) FL_Max: the maximum load force at the onset of maximum upward acceleration; (3) force ratio of FP_Peak to FL_Max; (4) percentage of maximal pinch strength: the FP_Peak divided by the maximal static pinch strength as a percentage of maximum voluntary contraction are detected in the initial evaluation.
The pinch-holding-up activity (PHUA) test | 6~8 weeks after intervention
  For the PHUA test, the participants were asked to pinch and lift the pinch device, and the pinch force will be recorded during the task. The raw force value would be collected and transferred into specific parameters include: (1) FP_Peak: the maximum pinch force during the lifting phase in the PHUA test; (2) FL_Max: the maximum load force at the onset of maximum upward acceleration; (3) force ratio of FP_Peak to FL_Max; (4) percentage of maximal pinch strength: the FP_Peak divided by the maximal static pinch strength as a percentage of maximum voluntary contraction are detected in the initial evaluation.
Semmes-Weinstein monofilament (SWM) | Baseline
  A touch-pressure threshold test with 20 nylon filaments with varying degrees of thickness is conducted. The examiner presses the filament at a 90° angle against the skin until it bows. When the patient indicates a response, the result is recorded. The filament is labeled with a numerical marking, which is a log to the base ten of the force in tenths of a milligram. The threshold value is the finest filament to which the subject correctly responds.
Semmes-Weinstein monofilament (SWM) | 6~8 weeks after intervention
  A touch-pressure threshold test with 20 nylon filaments with varying degrees of thickness is conducted. The examiner presses the filament at a 90° angle against the skin until it bows. When the patient indicates a response, the result is recorded. The filament is labeled with a numerical marking, which is a log to the base ten of the force in tenths of a milligram. The threshold value is the finest filament to which the subject correctly responds.
Purdue Pegboard test | Baseline
  The Purdue Pegboard test has high testing validity and reliability and has been broadly used to measure hand dexterity. The test comprises four subtests involving the ability of the subject to place pins in small holes with the dominant hand, non-dominant hand, and with both hands simultaneously, as well as performing an assembly task.
Purdue Pegboard test | 6~8 weeks after intervention
  The Purdue Pegboard test has high testing validity and reliability and has been broadly used to measure hand dexterity. The test comprises four subtests involving the ability of the subject to place pins in small holes with the dominant hand, non-dominant hand, and with both hands simultaneously, as well as performing an assembly task.
Michigan Hand Outcomes Questionnaire (MHQ) | Baseline
  Michigan Hand Outcomes Questionnaire (MHQ), a hand-specific outcomes instrument, is sensitive to providing an understanding of clinical changes with patients' self-reports. The MHQ contains six dimensions with 37 hand-specific questions. Higher scores indicate better hand function, with the exception of the pain facet. The testing reliability of MHQ ranges from 0.81 to 0.97.
Michigan Hand Outcomes Questionnaire (MHQ) | 6~8 weeks after intervention
  Michigan Hand Outcomes Questionnaire (MHQ), a hand-specific outcomes instrument, is sensitive to providing an understanding of clinical changes with patients' self-reports. The MHQ contains six dimensions with 37 hand-specific questions. Higher scores indicate better hand function, with the exception of the pain facet. The testing reliability of MHQ ranges from 0.81 to 0.97.
Diabetes-39 (D-39) | Baseline
  The Diabetes 39 (D-39) is a disease-specific questionnaire used to assess quality of life (QoL) in patients with diabetes. It contains of 39 questions regarding five dimensions, including energy and mobility, diabetes control, anxiety and worry, social and peer burden, and sexual functioning. Higher scores on all dimensions reveal a better QoL. The reliability of the Chinese version of the tool ranges from 0.82 to 0.93, and it also has good convergent and discriminant validity.
Diabetes-39 (D-39) | 6~8 weeks after intervention
  The Diabetes 39 (D-39) is a disease-specific questionnaire used to assess quality of life (QoL) in patients with diabetes. It contains of 39 questions regarding five dimensions, including energy and mobility, diabetes control, anxiety and worry, social and peer burden, and sexual functioning. Higher scores on all dimensions reveal a better QoL. The reliability of the Chinese version of the tool ranges from 0.82 to 0.93, and it also has good convergent and discriminant validity.
Moving two-point discrimination (M2PD) test | Baseline
  The Moving two-point discrimination test which is used to detect the shortest distance between the points that the subjects can perceive are tools for tactile acuity measuring. Also,it measures the innervation density of slowly and quickly adapting nerve fibers, respectively, and their corresponding mechanoreceptors as well.
Moving two-point discrimination (M2PD) test | 6~8 weeks after intervention
  The Moving two-point discrimination test which is used to detect the shortest distance between the points that the subjects can perceive are tools for tactile acuity measuring. Also,it measures the innervation density of slowly and quickly adapting nerve fibers, respectively, and their corresponding mechanoreceptors as well.
Static two-point discrimination (S2PD) test | Baseline
  The two-point discrimination test which is used to detect the shortest distance between the points that the subjects can perceive are tools for tactile acuity measuring.
Static two-point discrimination (S2PD) test | 6~8 weeks after intervention
  The two-point discrimination test which is used to detect the shortest distance between the points that the subjects can perceive are tools for tactile acuity measuring.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng-Kung University, Tainan, Taiwan